CLINICAL TRIAL: NCT07351760
Title: Outpatient Department Repair of Small Primary Ventral Hernias
Acronym: OPD-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPD-R
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Umbilical Hernia Repair; Epigastric Hernia Repair; Primary Ventral and Incisional Hernia Repair
Keywords: Local anesthesia; Hernia Repair; Daycare surgery; Umbilical hernia
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outpatient department repair (Experimental): Outpatient department repair of selected small primary ventral hernias under local anesthesia
  Interventions: Procedure: Outpatient department repair

INTERVENTIONS:
Procedure: Outpatient department repair — Outpatient department repair of selected small primary ventral hernias under local anesthesia

SUMMARY:
Ventral hernias are among the most common conditions requiring surgical intervention. Due to their benign nature, elective repairs of primary ventral hernias are usually given low priority for planned surgery. Routines for hernia repair that do not require operating theatre resources are therefore needed.

Repair under local anaesthesia has been demonstrated to be a safe and effective approach. While inguinal hernia repair under local anaesthesia is well established and extensively studied, primary ventral hernia repair under local anaesthesia has received comparatively limited attention. Although previous studies have demonstrated the safety of primary ventral hernias repair under local anaesthesia, most procedures are still performed in conventional operating theatres. The present prospective pilot study was therefore designed to assess the safety, feasibility, and patient satisfaction of repairing small, uncomplicated primary ventral hernias under local anaesthesia in the outpatient department using suture repair, without the resources available in the operating theatre.

The study is conducted as a single-arm pilot study. Adult patients of both sexes diagnosed with a small primary ventral hernia were assessed for eligibility. The primary outcome is the safety and feasibility of performing PVH repair under local anesthesia in the outpatient department, including patient tolerance and perioperative safety. Secondary outcomes included patient satisfaction, postoperative pain, and short-term recurrence.

Outpatient Department Repair is performed in a designated outpatient procedure room, separate from the conventional operating theatre. Local anesthesia is administered in a stepwise manner. Initially, local anesthesia is injected intradermally at the incision site. After confirming adequate anesthetic effect, a skin incision is made, and the subcutaneous tissue is dissected until the hernia sac is identified. Additional local anesthesia is applied directly into the wound at this stage.

For umbilical or paraumbilical hernias, the umbilicus is carefully separated from the hernia sac and surrounding fascia. During this phase, patients are asked standardized intraoperative questions while the surgeon continues the procedure. The hernia sac is reduced, and a further infiltration of local anesthesia is administered into the fascia adjacent to the defect.

The fascial defect is closed with a single horizontal running suture line using a continuous 2-0 polypropylene suture. When applicable, the umbilicus is reattached to the fascia using a 4-0 polydioxanone suture, positioned approximately 1 cm above or below the fascial suture line, to reduce the risk of suture sinus or chronic pain. The subcutaneous tissue is sutured with 3-0 polyglactin, and the skin is closed intracutaneously using 4-0 Monocryl.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Body mass index (BMI) ≤ 30 kg/m²
* Primary ventral hernia with fascia defect size < 2 cm

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Contraindications to local anaesthesia
* Pregnancy
* BMI > 30 kg/m²
* Ongoing anticoagulant therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Complications | 30 days
  Complications related to the procedure, including surgical site infections, hematoma and severe intraoperative pain

SECONDARY OUTCOMES:
Pain | Within two hours after surgery
  Intraoperative pain measured with visual analogue scale (VAS)
Hernia recurrence | Six months
  Hernia recurrence detected at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Karlskoga Hospital, Karlskoga, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Psuedonymized data are available on request from Gabriel Sandblom or Asmatullah Katawazai
Supporting Information: Study Protocol, SAP
Time Frame: January 2026 - December 2030
Access Criteria: Data are available on request to the responsible researchers.